CLINICAL TRIAL: NCT02184728
Title: Comparison of End-tidal Carbon Dioxide (ETCO2) Measured by Transportable Capnometer (EMMATM) and the Arterial pCO2 in General Anesthesia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Inje University (Other)
Responsible Party: Principal Investigator, Sira Bang, Assistant Professor, Inje University
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: IIT-2014-215
Record Dates: First submitted 2014-07-03; First posted 2014-07-09 (Estimated); Last update posted 2015-03-25 (Estimated); Status verified 2015-03

CONDITIONS: End Tidal Carbon Dioxide of Patients Undergoing General Anesthesia
Keywords: end-tidal CO2; capnometer

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- EMMA(TM) (No Intervention): A small capnograph for measuring ET-CO2 - the EMMA capnometer
  1
  Interventions: Device: End-tidal CO2(portable capnometer)

INTERVENTIONS:
Device: End-tidal CO2(portable capnometer) — End-tidal CO2(portable capnometer: EMMATM, Side stream capnometry module:Datex-Ohmeda S5 Anesthesia Monitor )levels were recorded at the time of arterial blood gas sampling.
  Other Names: EMMA(TM )

SUMMARY:
An end-tidal CO 2 monitor (capnometer) is used most often as a noninvasive substitute for PaCO2 in anesthesia, anesthetic recovery and intensive care. There is now also wide-spread use of capnometry on-site at emergency and trauma fields. So, portable device can be used usefully.

ELIGIBILITY:
Inclusion Criteria:

* patients who anticipated arterial gas analyze intraoperatively

Exclusion Criteria:

* patients who didn't get arterial line

Ages: 20 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2014-06; Primary Completion 2015-01 (Actual); Study Completion 2015-03 (Actual)

PRIMARY OUTCOMES:
End-tidal CO2 | During operation (2-4 times)
  End-tidal CO2(portable capnometer: EMMATM, Side stream capnometry module:Datex-Ohmeda S5 Anesthesia Monitor )levels were recorded at the time of arterial blood gas sampling.

CONTACTS AND LOCATIONS:
Locations (1):
- Inje University Seoul Paik Hospital, Seoul, Korea, Seoul, Jung-Gu,, South Korea

REFERENCES:
- [Derived] Kim KW, Choi HR, Bang SR, Lee JW. Comparison of end-tidal CO2 measured by transportable capnometer (EMMA capnograph) and arterial pCO2 in general anesthesia. J Clin Monit Comput. 2016 Oct;30(5):737-41. doi: 10.1007/s10877-015-9748-x. Epub 2015 Aug 12. PMID 26264607